CLINICAL TRIAL: NCT02742831
Title: A Theory-Based Intervention to Prevent Child Neglect in High-Risk
Brief Title: A Pilot Intervention With Families of Children With Special Health Care Needs
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects were enrolled and the grant period is ending.
Sponsor: Boston Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Caroline Kistin, BMC Attending Physician, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-35105; 1K23HD078503-01A1 (NIH)
Record Dates: First submitted 2016-04-05; First posted 2016-04-19 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Child Maltreatment; Children With Special Health Care Needs (CSHCN)
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive a one-on-one in-person intervention of 6 sessions, each lasting approximately 60 minutes. The intervention is intended to be delivered over a period of 12 weeks, with sessions occurring every 1-2 weeks. The overview of the 6 sessions is as follows:
  1. Behavioral chain analysis of episodes where parent felt stressed and episode where things went well. Identification of sources of interpersonal support.
  2. Stress relief. Development of a detailed crisis plan.
  3. Problem solving techniques.
  4. Emotional regulation exercises.
  5. Positive parenting, review of parenting challenges.
  6. Reflection, repeat behavioral chain analysis. Update crisis plan.
  Interventions: Behavioral: Intervention
- Control (Active Comparator): The families in the control group will be contacted by a member of the study team 6 times in 12 weeks to approximate the frequency of contact that the intervention group receives. The study team member will check in with families on the telephone or in person and will help them connect with clinic and community resources as needed.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Intervention — The intervention group will receive a 6-session intervention. The overview of the 6 sessions is as follows:
  1. "Behavioral chain analysis" of episode where parent felt stressed with child and episode where things went well. Identification of sources of interpersonal support.
  2. Stress relief techniques. Identification of short and long-term goals. Development of a detailed crisis plan.
  3. Problem solving techniques.
  4. Emotional regulation. Exercises to identify moods and explore connections between feelings, thoughts, and behavior.
  5. Positive parenting, review of common and specific parenting challenges, child development, short and long-term effects of different discipline approaches.
  6. Reflection, repeat behavioral chain analysis. Update crisis plan.
  Arms: Intervention
Other: Control — The families in the control group will be contacted by a member of the study team 6 times in 12 weeks to approximate the frequency of contact that the intervention group receives. The study team member will check in with families on the telephone or in person and will help them connect with clinic and community resources as needed.
  Arms: Control

SUMMARY:
This is a pilot randomized controlled trial of a behavioral intervention focused on improving parenting skills and preventing child neglect in families of children with special health care needs. The intervention focuses on problem solving, distress tolerance, and emotional regulation skills.

DETAILED DESCRIPTION:
This pilot randomized controlled trial will be conducted with 60 caregivers of children with special health care needs who have been reported to the child protection team at Boston Medical Center with concern for neglect that was ultimately not substantiated. Half of the subjects will be randomly assigned to receive the 6-session, one-on-one, in-person, behavioral intervention focused on problem solving, emotional regulation, and distress tolerance. The other half will be randomly assigned to the control group and will receive periodic check-ins and referrals to community resources as needed. Both groups will be followed for 12 months after randomization.

Children who have previously experienced neglect, or other forms of maltreatment, will not included in the study. Children will be defined as having special health care needs if they have a chronic physical, emotional, or behavioral condition.

With this pilot, the investigators aim to field-test study mechanics, including enrollment, randomization, and the collection of baseline and follow-up data; and obtain empiric estimates of study parameters to inform a subsequent fully-powered randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of a child under age 7 with a special health care need, defined as a chronic physical, emotional, or behavioral health condition
* Child has been referred to the Child Protection Team for neglect that was ultimately not substantiated
* Fluent in English or Spanish

Exclusion Criteria:

* Prior history of substantiated child maltreatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Study Logistics - subject enrollment | Monthly change from baseline to 12 months post randomization
  As this is a pilot study, the primary objective is to field test study logistics, including subject enrollment. The investigators will review monthly counts of enrolled subjects from baseline to 12 months post-randomization, and will compare the number of subjects in each study arm to target enrollment goals. Because of emerging consensus that group-to-group comparisons in a pilot study are not only invalid but also misleading, estimating effect size is deliberately not our primary study objective.
Study Logistics - fidelity of intervention delivery | 3 months post randomization
  For the intervention group, treatment fidelity will be assessed by audio taping a random 10% of sessions and scoring them with standardized instruments. The investigators will measure the proportion of sessions delivered with fidelity. Because of emerging consensus that group-to-group comparisons in a pilot study are not only invalid but also misleading, estimating effect size is deliberately not our primary study objective.

SECONDARY OUTCOMES:
Re-referral to child protection team or social services | 3 months post randomization
  The investigators will obtain empirical estimates of the proportion of control group subjects to be re-referred to child protection team or social services by 3 months post randomization. This will allow the investigators to power a later study for this dichotomous outcome.
Re-referral to child protection team or social services | 6 months post randomization
  The investigators will obtain empirical estimates of the proportion of control group subjects to be re-referred to child protection team or social services by 6 months post randomization. This will allow the investigators to power a later study for this dichotomous outcome.
Re-referral to child protection team or social services | 12 months post randomization
  The investigators will obtain empirical estimates of the proportion of control group subjects to be re-referred to child protection team or social services by 12 months post randomization. This will allow the investigators to power a later study for this dichotomous outcome.
Adherence to recommended medical care | 3 months post randomization
  The investigators will conduct chart review to count the number of missed medical appointments, emergency department visits, and hospitalizations in the 90 days preceding the analysis. The investigators will specifically examine the proportion of control group subjects to experience each outcome and will use this data to power a later study.
Adherence to recommended medical care | 6 months post randomization
  The investigators will conduct chart review to count the number of missed medical appointments, emergency department visits, and hospitalizations in the 90 days preceding the analysis. The investigators will specifically examine the proportion of control group subjects to experience each outcome and will use this data to power a later study.
Adherence to recommended medical care | 12 months post randomization
  The investigators will conduct chart review to count the number of missed medical appointments, emergency department visits, and hospitalizations in the 90 days preceding the analysis. The investigators will specifically examine the proportion of control group subjects to experience each outcome and will use this data to power a later study.

OTHER OUTCOMES:
Parental well-being and mental health - Quick Inventory of Depressive Symptomatology | Change in score from baseline to 12 months post randomization
  The investigators will use validated measures to evaluate parental well-being. The measures include the Quick Inventory of Depressive Symptomatology. The investigators will analyze the measure as a continuous variable (overall score) and dichotomous variable (depression present or absent) and will obtain empirical estimates of the following study parameters to inform power calculations for a subsequent study: 1) within-group standard deviation of each continuous outcome measure; 2) proportion of control group subjects to experience each dichotomous outcome; and 3) correlation over time of the outcome measured at both baseline and follow-up. This will allow the investigators to power a later study, for both dichotomous and continuous outcomes.
Parental well-being and mental health - the Social Adjustment Scale-Short Report | Change in score from baseline to 12 months post randomization
  The investigators will use validated measures to evaluate parental well-being. The measures include the Social Adjustment Scale-Short Report. The investigators will analyze the measure as a continuous variable (overall score) and dichotomous variable (social adjustment present or absent) and will obtain empirical estimates of the following study parameters to inform power calculations for a subsequent study: 1) within-group standard deviation of each continuous outcome measure; 2) proportion of control group subjects to experience each dichotomous outcome; and 3) correlation over time of the outcome measured at both baseline and follow-up. This will allow the investigators to power a later study, for both dichotomous and continuous outcomes.
Parental well-being and mental health - the Medical Outcomes Survey Social Support | Change in score from baseline to 12 months post randomization
  The investigators will use validated measures to evaluate parental well-being. The measures include the Medical Outcomes Survey Social Support. The investigators will analyze the measure as a continuous variable (overall score) and dichotomous variable (social support present or absent) and will obtain empirical estimates of the following study parameters to inform power calculations for a subsequent study: 1) within-group standard deviation of each continuous outcome measure; 2) proportion of control group subjects to experience each dichotomous outcome; and 3) correlation over time of the outcome measured at both baseline and follow-up. This will allow the investigators to power a later study, for both dichotomous and continuous outcomes.
Parental well-being and mental health - the Perceived Stress Scale | Change in score from baseline to 12 months post randomization
  The investigators will use validated measures to evaluate parental well-being. The measures include the Perceived Stress Scale. The investigators will analyze the measure as a continuous variable (overall score) and dichotomous variable (stress present or absent) and will obtain empirical estimates of the following study parameters to inform power calculations for a subsequent study: 1) within-group standard deviation of each continuous outcome measure; 2) proportion of control group subjects to experience each dichotomous outcome; and 3) correlation over time of the outcome measured at both baseline and follow-up. This will allow the investigators to power a later study, for both dichotomous and continuous outcomes.
Parental well-being and mental health - the Parenting Stress-Short Form | Change in score from baseline to 12 months post randomization
  The investigators will use validated measures to evaluate parental well-being. The measures include the Parenting Stress-Short Form. The investigators will analyze the measure as a continuous variable (overall score) and dichotomous variable (parenting stress present or absent) and will obtain empirical estimates of the following study parameters to inform power calculations for a subsequent study: 1) within-group standard deviation of each continuous outcome measure; 2) proportion of control group subjects to experience each dichotomous outcome; and 3) correlation over time of the outcome measured at both baseline and follow-up. This will allow the investigators to power a later study, for both dichotomous and continuous outcomes.
Parental well-being and mental health - the Parenting Scale | Change in score from baseline to 12 months post randomization
  The investigators will use validated measures to evaluate parental well-being. The measures include the Parenting Scale. The investigators will analyze the measure as a continuous variable (overall score) and dichotomous variable (parenting style present or absent) and will obtain empirical estimates of the following study parameters to inform power calculations for a subsequent study: 1) within-group standard deviation of each continuous outcome measure; 2) proportion of control group subjects to experience each dichotomous outcome; and 3) correlation over time of the outcome measured at both baseline and follow-up. This will allow the investigators to power a later study, for both dichotomous and continuous outcomes.
Parental well-being and mental health - the Parent Development Interview-Revised | Change in score from baseline to 12 months post randomization
  The investigators will use validated measures to evaluate parental well-being. The measures include the Parent Development Interview-Revised. The investigators will analyze the measure as a continuous variable (overall score) and dichotomous variable (reflective functioning present or absent) and will obtain empirical estimates of the following study parameters to inform power calculations for a subsequent study: 1) within-group standard deviation of each continuous outcome measure; 2) proportion of control group subjects to experience each dichotomous outcome; and 3) correlation over time of the outcome measured at both baseline and follow-up. This will allow the investigators to power a later study, for both dichotomous and continuous outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline J Kistin, MD, MSc, Principal Investigator — Boston University School of Medicine/Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No